CLINICAL TRIAL: NCT00728299
Title: The Effects of Consumption of Pomegranate Juice on Carotid Intima-Media Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiant Research (Other)
Collaborators: Roll International Corporation (Industry)
Responsible Party: Michael H. Davidson, MD, Executive Medical Director,, Radiant Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Radiant Development #202528
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease, carotid intima-media thickness
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PomWonderful Juice
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo juice

INTERVENTIONS:
Drug: PomWonderful Juice — 8 oz per day each day for 78 weeks
  Arms: 1
Drug: Placebo juice — 8 oz per day for 78 weeks
  Arms: 2

SUMMARY:
Increases in carotid artery intima-media thickness (IMT) are correlated with increased risk of stroke and myocardial infarction. The purpose of this study is to assess if pomegranate juice will retard the carotid (IMT) progression rate in men and women who have one or more existing cardiovascular risk factors (current cigarette smoking, hypertension, low HDL-cholesterol, and/or high LDL-cholesterol) upon entrance into the study.

DETAILED DESCRIPTION:
Previous studies in atherosclerotic mice have shown that pomegranate supplementation reduced their macrophage oxidative stress and attenuated the development of their atherosclerosis. Further research in hypertensive humans demonstrated that pomegranate juice had an angiotensin converting enzyme (ACE)-inhibitory effect and significantly decreased systolic blood pressure.

This study will use a randomized, double-blind, placebo-controlled design with eight clinic visits (one screening visit [week -4 to -1], one baseline visit [week 0], and six treatment visits [weeks 13, 26, 38, 52, 65, and 78]).

ELIGIBILITY:
Inclusion Criteria:

* Males between the ages of 45 and 74 and females between the ages of 55 and 74 years.
* Subject has ≥ 1 of the following risk factors at Visit 1 (week -4 to -1):

  * current cigarette smoking (defined as any cigarette smoking within the past month)
  * hypertension (blood pressure ≥ 140/90 mm Hg or using an antihypertensive medication)
  * low HDL cholesterol (< 40 mg/dL)
  * high LDL cholesterol (≥ 130 mg/dL and < 190 mg/dL), on statin therapy or not
* Posterior wall common carotid IMT > 0.7 mm and < 2.0 mm at Visit 2 (week 0) with an adequate image on at least one side.
* Subject understands the study procedures and signs an informed consent form.
* Normally active and judged to be in good health on the basis of medical history, physical examination, and routine laboratory tests.

Exclusion Criteria:

* Use of any pharmacologic lipid-altering medications, besides statins (e.g., fibrate derivatives, bile acid binding resins, and niacin or its analogues at doses > 400 mg/d) six weeks prior to Visit 1
* Body mass index > 40 kg/m2.
* Unstable use (< 2 months prior to Visit 1) of any supplement known to alter lipid metabolism, including but not limited to: dietary fiber supplements (including > 2 teaspoons Metamucil® or psyllium-containing supplement per day), omega-3 fatty acid supplements, sterol/stanol products, red rice yeast supplements, garlic supplements, soy isoflavone supplements or others at the discretion of the Investigator).
* History of pomegranate consumption (either eating pomegranates or drinking pomegranate juice) within the past 6 months.
* Clinical evidence or history of coronary heart disease (CHD) or CHD equivalents including:

  * diabetes mellitus,
  * angina,
  * myocardial infarction,
  * transient ischemic attack,
  * symptomatic carotid artery disease,
  * cerebrovascular accident,
  * coronary artery bypass grafting,
  * percutaneous transluminal coronary angioplasty,
  * peripheral arterial disease,
  * abdominal aortic aneurysm,
  * ankle brachial index < 0.90,
  * and/or a Framingham Risk Score ≥ 16 points for men and ≥ 23 points for women (10-year CHD risk > 20%)
* Active cancer, other than non-melanoma skin cancer, within the previous two years.
* Prior diagnosis of human immunodeficiency virus (HIV) or hepatitis B or hepatitis C.
* Uncontrolled hypertension (average systolic blood pressure ≥ 160 mm Hg and/or average diastolic blood pressure ≥ 100 mm Hg).
* Untreated or unstable hypothyroidism (receiving stable dose therapy for < 4.0 months).
* Concomitant use of beta-adrenergic blockers or immunosuppressants
* Concomitant use of estrogen or progestin therapy.
* Allergy to pomegranates or pomegranate juice.
* Known allergy to blood products.
* Non-English speaking.
* Active liver disease or hepatic dysfunction as defined by elevations of ≥ 2.0 x ULN at Visit 1 in any of the following liver function tests: ALT, AST or bilirubin.
* Serum creatinine > 2.0 mg/dL recorded during screening period.
* Recent history of (within past 12 months) or strong potential for alcohol or substance abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 4 oz wine, or 1 ½ oz distilled spirits).
* Participation in another clinical study within 30 days prior to screening visit 1 (week -4 to -1).
* Has a condition the Investigator believes would interfere with evaluation of the subject, or may put subject at undue risk.
* Posterior wall common carotid IMT ≥ 2.0 mm on either side at Visit 2 (week 0).

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2003-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Difference in posterior wall common carotid intima-media thickness (IMT) progression rate in mm/yr between PomWonderful juice and placebo, utilizing non-contrast images | 78-90 weeks

SECONDARY OUTCOMES:
Difference between placebo and PomWonderful juice in internal carotid artery IMT progression rate in mm/yr | 78-90 weeks
Difference between placebo and PomWonderful juice in the carotid bifurcation IMT progression rate in mm/yr | 78-90 weeks
Difference between placebo and PomWonderful juice in the anterior wall common carotid IMT progression rate in mm/yr, without contrast agent | 78-90 weeks
Difference between placebo and PomWonderful juice in the anterior wall common carotid IMT progression rate in mm/yr, with contrast agent | 78-90 weeks
Difference between placebo and PomWonderful juice in the posterior wall common carotid IMT progression rate in mm/yr, with contrast agent | 78-90 weeks
Difference between placebo and PomWonderful juice in the composite IMT measure, which combines the measurements of the common and internal carotid and the carotid bifurcation in mm/yr | 78-90 weeks
Change from baseline to 13 weeks in hs-CRP concentration | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD, Principal Investigator — FACC